CLINICAL TRIAL: NCT05351788
Title: A Phase Ⅱ Clinical Study of Combination Therapy of SKB264 in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: SKB264 Combinatiton Therapy in Patients With Advanced or Metastatic Non-small Cell Lung Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅱ-05
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 18-O-demethylcervinomycin A2; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SKB264+KL-A167 (Experimental): Participants received SKB264 followed by KL-A167
  Interventions: Drug: SKB264; Drug: KL-A167
- SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR wide type) (Experimental): Participants received SKB264 followed by KL-A167 with Carboplatin or Cisplatin
  Interventions: Drug: SKB264; Drug: KL-A167; Drug: Carboplatin; Drug: Cisplatin
- SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR mutation) (Experimental): Participants received SKB264 followed by KL-A167 with Carboplatin or Cisplatin
  Interventions: Drug: SKB264; Drug: KL-A167; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: SKB264 — SKB264 will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle (5mg/kg)
Drug: KL-A167 — KL-A167 will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle (1200mg Q3W)
Drug: Carboplatin — Carboplatin will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle（AUC 5)
  Arms: SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR mutation); SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR wide type)
Drug: Cisplatin — Cisplatin will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle (75mg/m²)
  Arms: SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR mutation); SKB264+KL-A167+ Carboplatin or Cisplatin (EGFR wide type)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary antitumor activity of SKB264 in combination with KL-A167 with or without chemotherapy with advanced or metastatic non-small cell lung cancer. The study is divided into two parts. Part 1 will be the safety run-in phase, and Part 2 will be the cohort expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 and ≤ 75 years of age at the time of signing the informed consent form;
2. Histologically and cytologically confirmed NSCLC;
3. Cohort 1: Patients with locally advanced/metastatic NSCLC with wild-type EGFR and negative ALK fusion gene, no or at most one prior line of systemic chemotherapy regimen for advanced or metastatic NSCLC. Cohort 2: Patients with locally advanced/metastatic NSCLC with wild-type EGFR and negative ALK fusion gene, no prior systemic therapy. Cohort 3: Patients with locally advanced/metastatic NSCLC with EGFR activating mutation and negative ALK fusion gene, who have failed previous treatment with EGFR-TKIs.
4. Provide fresh or archival tumor tissue for biomarker testing and analysis;
5. Patients with at least one measurable lesion per RECIST v1.1 criteria, and patients with only skin or bone lesions cannot be enrolled;
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with an expected survival of ≥ 12 weeks;
7. Adequate organ and bone marrow function
8. For female patients of childbearing age and male patients with partners of childbearing age, they must use effective medical contraception during the study treatment period and for 6 months after the last dose of study medication (see Annex for specific contraceptive measures);
9. Each patient must voluntarily agree to participate in the study, sign the informed consent form, and comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Presence of small cell lung carcinoma (SCLC) components in histological pathology;
2. History of other malignancies;
3. Presence of metastases to brainstem, meninges and spinal cord, or spinal cord compression;
4. Presence of active central nervous system (CNS) metastases;
5. Imaging (CT or MRI) shows that the tumor surrounds important blood vessels, or the investigator determines that the tumor is most likely to invade important blood vessels during the subsequent study to cause fatal major hemorrhage;
6. Serious or uncontrolled cardiac disease or clinical symptoms requiring treatment, including any of the following:
7. Patients with (noninfectious) interstitial lung disease (ILD) or history of pneumonia requiring steroid therapy; patients with serious pulmonary function impairment due to lung disease;
8. Uncontrolled systemic disease as judged by the investigator, included uncontrolled hypertension, uncontrolled diabetes, pesence of pleural effusion, pericardial effusion, or ascites that is clinically symptomatic or requires repeated drainage;
9. Certain viral infections including active hepatitis B or hepatitis C; known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); or positive syphilis antibody test;
10. Known active tuberculosis;
11. Known hypersensitivity to the study drug or any of its components, or severe allergic reactions to other monoclonal antibodies;
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Pregnant or lactating women;
14. Any patient whose condition deteriorates rapidly during the screening process prior to the first dose, such as severe changes in performance status, unstable pain requiring adjustment of analgesic therapy, etc
15. Other circumstances that, in the opinion of the investigator, are not appropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From baseline up to 30 days after last dose or to the beginning of the new anti-cancer therapy, up to 24 months
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Objective Response Rate (ORR) | From baseline to first documented objective response, up to 24 months
  Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Investigator based on RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From baseline to the first documented disease progression or date of death (whichever occurs first), up to 24 months
  Progression-free survival (PFS) was defined as the time from baseline to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions.
Duration of response (DOR) | From the date of first objective response (CR or PR) to the date of first documentation of PD or death (whichever occurs first), up to 24 months
  Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR was measured for responding subjects (PR or CR) only.
Disease control rate (DCR) | From baseline to date of first documented objective response (CR, PR, and SD), up to 24 months
  Disease control rate (DCR) was defined as the sum of complete response (CR) rate, partial response (PR) rate, and stable disease (SD) rate. As per RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of SKB264-ADC, SKB264-TAB and free KL610023 | Cycle 1-8, every 4 cycles starting from Cycle 12 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months
Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of SKB264-ADC, SKB264-TAB and free KL610023 | Cycle 1-8, every 4 cycles starting from Cycle 12 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of KL-A167 | Cycle 1-8, every 4 cycles starting from Cycle 12 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months
Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of KL-A167 | Cycle 1-8, every 4 cycles starting from Cycle 12 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months
Anti-drug Antibodies (ADA) for SKB264 and KL-A167 | Cycle 1-8, every 4 cycles starting from Cycle 12 Day 1: pre-dose, post-dose (each cycle is 21 days), up to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou

REFERENCES:
- [Derived] Hong S, Wang Q, Cheng Y, Luo Y, Qu X, Zhu H, Ding Z, Li X, Wu L, Wang Y, Hu S, Wang E, Liu A, Sun Y, Fan Y, Ye F, Lu K, Fang J, Shen Y, Jin X, Ge J, Zhang L, Fang W. First-line sacituzumab tirumotecan with tagitanlimab in advanced non-small-cell lung cancer: a phase 2 trial. Nat Med. 2025 Nov;31(11):3654-3661. doi: 10.1038/s41591-025-03883-5. Epub 2025 Aug 19. PMID 40830660